CLINICAL TRIAL: NCT03208582
Title: Do Bisphosphonates Alter the Skeletal Response to Mechanical Stimulation in Children With Osteogenesis Imperfecta?
Acronym: BAMES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SCH-2013
Record Dates: First submitted 2017-05-23; First posted 2017-07-05 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2017-05

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Risedronic Acid; Diphosphonates; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm trial (Other): Intervention : Risedronate Sodium (oral) Dosage: 1mg/kg/week Frequency: once/week Duration: 6 weeks
  Interventions: Drug: Risedronate Sodium; Dietary Supplement: Calcichew tablets

INTERVENTIONS:
Drug: Risedronate Sodium — Participants will be initially tested on the response to mechanical stimulation as a baseline and then tested again after 6 weeks treatment with Risedronate
  Other Names: Bisphosphonate
Dietary Supplement: Calcichew tablets — Participants will take calcichew tablets during the 6 week period of risedronate treatment

SUMMARY:
Osteogenesis Imperfecta(OI) is an inherited disorder characterised by extreme fragility of the bones. Bones often break from little or no apparent cause.

Current available medicine can increase bone strength by making bones wider and "filling in" the holes in the bone walls that weaken it. These medicines are bisphosphonates, given either by a drip intravenously (eg pamidronate), or taken by mouth (eg risedronate). Their major action is to prevent bone breakdown by stopping the normal process of removing and then replacing old bone tissue, so in some parts of the bone, new bone formation is actually reduced. Most studies of bisphosphonates in children with OI have shown increased bone mineral density and improved exercise tolerance that could positively affect new bone formation; some have shown reduced fracture rate. Bone is highly responsive to mechanical stimulation. Whole body vibration (WBV) is a form of mechanical stimulation that has been shown to improve bone mineral density in some individuals with narrow bones.

Little is known whether bisphosphonates affect the response of the skeleton to mechanical stimulation. We will determine the response to mechanical stimulation in children with OI by looking at bone turnover markers following WBV in those who are and are not treated with bisphosphonates.

The results from this study will help us to understand whether skeleton in children with OI is normally responsive to mechanical stimulation, and whether bisphosphonates alter that responsiveness in a way that is either beneficial or not for increasing bone strength.

DETAILED DESCRIPTION:
Essentially, subjects will have a baseline assessment (WBV1) of their bone turnover marker response to a week-long period of whole body vibration (10 minutes/day), followed by a "washout period" of 5 weeks during which bone turnover is expected to return to normal. Following this, there will be a period of 6 weeks of treatment with risedronate (1 mg/kg/week). Immediately following this will come a second assessment (WBV2) of the bone turnover marker response to a week-long period of whole body vibration (10 minutes/day) as previously.

The subjects stand on the vibration platform for 10 minutes for 7 days on 2 occasions. The vibration is delivered as 4 "blocks" of 2.5 minutes each, with 30 seconds rest in between each block. The initial Whole Body Vibration (WBV) on day 1 will be undertaken in the Sheffield Children's Hospital Clinical Research Facility (SCHCRF) under supervision. Subsequent WBVs D2-D7 and D85-91 will be done in the participants' homes. Participants will be asked to record the administration and timing of WBV in a diary.

Blood samples will be taken after an overnight fast according to the following schedule:

Pre-WBV1 D1; D8 (postWBV); D15; D43 (immediate pre-risedronate); D85 (post-risedronate and pre-WBV2); D92 (post-WBV2) and D99 (final). 7 samples are taken altogether.

The blood tests are bone turnover markers (Alkaline phosphatase[ALP], Procollagen Type 1 N-Terminal Propeptide[P1NP] and C-Terminal Telopeptide of Type 1 Collagen[CTX]). The first blood test will be done by the researcher (Dr Sithambaram) in the SCHCRF and the subsequent 6 blood tests can be done by the research nurse/researcher at the participant's home. Blood samples taken will be allowed to clot for ½ an hour. Samples will be spun at 2500 rpm for 10 minutes at 4°C. The centrifuged sample will be stored in SCHCRF at -80°C. Blood tests will be analysed in the Mellanby Centre for Bone Research, University of Sheffield.

Participants will be taking risedronate (oral bisphosphonate, once weekly), rounded to the nearest 5 mg) together with Vitamin D and calcium for 6 weeks. Vitamin D and Calcium will be given as Calcichew 500mg/200 IU tablets, 1 tablet for participants weighing less than 30 kg and 2 tablets for participants weighing 30 kg or more. Risedronate Sodium belongs to Bisphosphonates group of medicine. As per BNF, it is not licensed for use in children. The trade name is Actonel® Warner Chilcott). This study will use 5mg and 35mg film-coated tablets.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-16 years
* Able to speak fluent English
* Diagnosed with osteogenesis imperfecta
* Able to stand
* Not treated with bisphosphonates

Exclusion Criteria:

* Presence of other chronic illnesses
* Balance problems
* Recent fracture (in the last 6 months)
* Recent (last 12 months) or current treatment likely to affect bone - this does not include inhaled or intermittent oral therapy with steroids for asthma
* Involvement in another interventional research project

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Change in P1NP response to 1 week of vibration without risedronate treatment, followed by a washout period. Change in P1NP response to vibration will be reassessed following Risedonate treatment. Serial bone markers will be done over a 99 day period. | 99 days
  To assess if risedronate alters the response to mechanical stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bishop, MD, FRCPCH, Study Chair — Sheffield Children's Hospital and University of Sheffield
Locations (1):
- Clinical Research Facility, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided